CLINICAL TRIAL: NCT01527630
Title: A Randomised, Double-blind, Single-centre, Two-Period Crossover Trial Testing the Bioequivalence of Two Formulations of NN-X14Mix50 in Healthy Japanese Subjects
Brief Title: Bioequivalence of Two Formulations of Biphasic Insulin Aspart 50 in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIASP-1504
Record Dates: First submitted 2012-02-02; First posted 2012-02-07 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formulation A (Experimental)
  Interventions: Drug: biphasic insulin aspart 50
- Formulation B (Experimental)
  Interventions: Drug: biphasic insulin aspart 50

INTERVENTIONS:
Drug: biphasic insulin aspart 50 — A single dose of each formulation administered subcutaneously (s.c., under the skin) on 2 dosing visits separated by a wash-out period of 6-21days

SUMMARY:
This trial is conducted in Japan. The aim of this trial is to investigate the bioequivalence of two formulations of biphasic insulin aspart 50 (NN-X14Mix50) in healthy Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Considered generally healthy upon completion of medical history and physical examination, as judged by the Investigator or Sub-Investigator.
* Body Mass Index (BMI) between 19-29 kg/m^2 (inclusive)
* Fasting plasma glucose between 3.8-6.0 mmol/L (both inclusive)

Exclusion Criteria:

* Clinically significant abnormal haematology, biochemistry or urinalysis screening tests, as judged by the Investigator or Sub-Investigator
* Any serious systemic infectious disease that had occurred during the 4 weeks prior to the screening, as judged by the Investigator or Sub-Investigator
* Any inter-current illness that might affect blood glucose, as judged by the Investigator or Sub-Investigator
* Hepatitis B or C, or HIV (human immunodeficiency virus) positive
* Subjects with a first degree relative with diabetes mellitus
* History of or presence of diabetes, cancer or any clinically significant cardiac, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, dermatological, venereal, haematologic, neurologic, or psychiatric diseases or disorder
* Subjects who consumed more than 28 units of alcohol per week or who had a significant history of alcoholism or drug/chemical abuse
* Subjects who smoked more than 5 cigarettes per day
* Subjects who had taken part in strenuous exercise within 7 days prior to the screening

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2002-11-16 (Actual); Primary Completion 2003-01-08 (Actual); Study Completion 2003-01-08 (Actual)

PRIMARY OUTCOMES:
Area under the insulin aspart concentration-time curve in the interval from 0 to 16 hours
Cmax, maximum insulin aspart concentration

SECONDARY OUTCOMES:
Area under the insulin aspart concentration-time curve
Tmax, time to maximum insulin aspart concentration
MRT, mean residence time
t½, terminal half-life

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com